CLINICAL TRIAL: NCT00685113
Title: A Multicenter, Randomized, Double-Blind, Parallel Group Study to Evaluate the Efficacy and Safety of Two Doses of DR-3001 Versus Placebo in Women With Overactive Bladder
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of DR-3001 in Women With Overactive Bladder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duramed Research (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DR-OXY-301
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: DR-3001
- 2 (Experimental)
  Interventions: Drug: DR-3001
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DR-3001 — 4mg/day vaginal ring inserted vaginally and replaced every 4 weeks
  Other Names: Oxybutinyn Vaginal Ring
  Arms: 1
Drug: DR-3001 — 6mg/day vaginal ring inserted vaginally and replaced every 4 weeks
  Other Names: Oxybutinyn Vaginal Ring
  Arms: 2
Drug: Placebo — Placebo vaginal ring inserted vaginally and replaced every 4 weeks
  Arms: 3

SUMMARY:
This is a multicenter study to evaluate the efficacy and safety of 2 different doses of DR-3001. For eligible subjects the duration of the study will be approximately 20 weeks; this will consist of a 4-week screening period, a 12-week treatment period and a 4-week follow-up period. Subjects will have physical and laboratory exams, including blood draws at each scheduled visit. Subjects will be required to insert a vaginal ring (replacing it every 4 weeks) and to keep a daily record of their toilet voids (including time,type and volume) for 3 days at several specified time points.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age or older, ambulatory, with a history and presentation consistent with urge incontinence ≥ 6 months
* Able to distinguish between stress and urge incontinence
* During the Screening Period able to demonstrate the presence of overactive bladder with urge incontinence based on diary entries
* Others as dictated by FDA-approved protocol

Exclusion Criteria:

* Stress incontinence, continuous incontinence or overflow urinary incontinence
* Chronic illness, neurological dysfunction or injury that could cause incontinence
* Pregnant, breastfeeding, or gave birth in the last 6 months
* Others as dictated by FDA-approved protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1104 (Actual)
Dates: Start 2008-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Change in total weekly number of incontinence (urge and stress)episodes | Baseline to end-of-treamtent (Week 12/Early withdrawal)

SECONDARY OUTCOMES:
Change in average daily urinary frequency and average void volume | Baseline to end-of-treamtent (Week 12/Early withdrawal)
Proportion of subjects with no incontinence episodes recorded in the final 3-day diary | Final 3-day diary
3 subject-reported outcome measures: visual analogue scale of OAB symptoms, Urogenital Distress Inventory, Incontinence Impact Question | Baseline to end-of-treatment (Week 12/Early Withdrawal)
Adverse events (AEs) reported by subjects or identified by the investigator | Basline to end-of-treatment (Week 12/Early Withdrawal)

CONTACTS AND LOCATIONS:
Overall Officials: Duramed Research Protocol Chair, Study Chair — Duramed Research, Inc.
Locations (74):
- United States (71):
  - Duramed Investigational Site, Huntsville, Alabama
  - Duramed Investigational Site, Mobile, Alabama
  - Duramed Investigational Site, Montgomery, Alabama
  - Duramed Investigational Site, Phoenix, Arizona
  - Duramed Investigational Site, Tucson, Arizona
  - Duramed Investigational Site, Little Rock, Arkansas
  - Duramed Investigational Site, Encinitas, California
  - Duramed Investigational Site, Los Angeles, California
  - Duramed Investigational Site, San Diego, California
  - Duramed Investigational Site, Colorado Springs, Colorado
  - Duramed Investigational Site, Denver, Colorado
  - Duramed Investigational Site, Danbury, Connecticut
  - Duramed Investigational Site, Milford, Connecticut
  - Duramed Investigational Site, New London, Connecticut
  - Duramed Investigational Site, Aventura, Florida
  - Duramed Investigational Site, Gainesville, Florida
  - Duramed Investigational Site, Jacksonville, Florida
  - Duramed Investigational Site, Miami, Florida
  - Duramed Investigational Site, New Port Richey, Florida
  - Duramed Investigational Site, Tampa, Florida
  - Duramed Investigational Site, West Palm Beach, Florida
  - Duramed Investigational Site, Atlanta, Georgia
  - Duramed Investigational Site, Augusta, Georgia
  - Duramed Investigation Site, Decatur, Georgia
  - Duramed Investigational Site, Savannah, Georgia
  - Duramed Investigational Site, Boise, Idaho
  - Duramed Investigational Site, Coeur d'Alene, Idaho
  - Duramed Investigational Site, Meridian, Idaho
  - Duramed Investigational Site, Fort Wayne, Indiana
  - Duramed Investigational Site, Jeffersonville, Indiana
  - Duramed Investigational Site, South Bend, Indiana
  - Duramed Investigational Site, Newton, Kansas
  - Duramed Investigational Site, Wichita, Kansas
  - Duramed Investigational Site, Louisville, Kentucky
  - Duramed Investigational Site, Lafayette, Louisiana
  - Duramed Investigational Site, Marrero, Louisiana
  - Duramed Investigational Site, Shreveport, Louisiana
  - Duramed Investigational Site, Watertown, Massachusetts
  - Duramed Investigational Site, Las Vegas, Nevada
  - Duramed Investigational Site, North Las Vegas, Nevada
  - Duramed Investigational Site, Lebanon, New Hampshire
  - Duramed Investigational Site, Lawrenceville, New Jersey
  - Duramed Investigational Site, Moorestown, New Jersey
  - Duramed Investigational Site, New Brunswick, New Jersey
  - Duramed Investigational Site, Albuquerque, New Mexico
  - Duramed Investigational Site, Port Jefferson, New York
  - Duramed Investigational Site, New Bern, North Carolina
  - Duramed Investigational Site, Winston-Salem, North Carolina
  - Duramed Investigational Site, Cleveland, Ohio
  - Duramed Investigational Site, Mayfield Heights, Ohio
  - Duramed Investigational Site, Bethany, Oklahoma
  - Duramed Investigational Site, Oklahoma City, Oklahoma
  - Duramed Investigational Site, Eugene, Oregon
  - Duramed Investigational Site, Medford, Oregon
  - Duramed Investigational Site, Philadelphia, Pennsylvania
  - Duramed Investigational Site, Pittsburgh, Pennsylvania
  - Duramed Investigational Site, Pottstown, Pennsylvania
  - Duramed Investigational Site, Charlestown, South Carolina
  - Duramed Investigational Site, Columbia, South Carolina
  - Duramed Investigational Site, Greensville, South Carolina
  - Duramed Investigational Site, Hilton Head Island, South Carolina
  - Duramed Investigational Site, Jackson, Tennessee
  - Duramed Investigational Site, Dallas, Texas
  - Duramed Investigational Site, Houston, Texas
  - Duramed Investigational Site, San Antonio, Texas
  - Duramed Investigational Site, Waco, Texas
  - Duramed Investigational Site, Salt Lake City, Utah
  - Duramed Investigational Site, Williston, Vermont
  - Duramed Investigational Site, Norfolk, Virginia
  - Duramed Investigational Site, Seattle, Washington
  - Duramed Investigational Site, Tacoma, Washington
- Canada (3):
  - Duramed Investigatinal Site, Vancouver, British Columbia
  - Duramed Investigational Site, Oshawa, Ontario
  - Duramed Investigational Site, Thunder Bay, Ontario